CLINICAL TRIAL: NCT03826095
Title: Investigation of the Effects of Respiratory Functions and Trunk Control on Functional Mobility in Individuals With Multiple Sclerosis
Brief Title: Respiratory Functions, Trunk Control and Mobility Evaluation in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: KARMUTLU (Unknown); MATUNCER (Unknown); EÇKÜTÜKÇÜ (Unknown)
Responsible Party: Principal Investigator, MELIKE SUMEYYE CENGIZ, Principal Investigator, Hacettepe University
Other Study IDs: Assesment in MS
Record Dates: First submitted 2019-01-23; First posted 2019-02-01 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Physical Therapy
Keywords: Multiple Sclerosis; Respiratory function; Respiratory muscle strength; Trunk control; Functional mobility
MeSH Terms: conditions — Multiple Sclerosis; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple Sclerosis: Patients with a clinically definitive diagnosis of MS, 0-5.5 Extended Disability Status Scale range.
- Healthy individuals: Voluntary healthy individuals with similar age and gender

SUMMARY:
Respiratory functions and body control are affected in patients with multiple sclerosis (MS). Because of this effect, the dependency of individuals increases in daily living activities and their quality of life decreases.

We think that respiratory functions, respiratory muscle strength and trunk control affect vital mobility as well as vital importance for individuals with MS. As a result of the investigations, it is concluded that the literature is insufficient in this area.

The aim of this study is to investigate the effects of pulmonary function, respiratory muscle strength and trunk control on functional mobility in individuals with MS and compare with healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Having a definite MS diagnosis
* Up to 5.5 points on the Scored Disability Status Scale (EDSS)
* In the last 3 months have not experienced an attack
* Mini mental test score of 24 and above
* Acceptance to participate in the study.

Exclusion Criteria:

* Having orthopedic problems
* The presence of other neurological problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MS patients who are ambulatory
  Healthy volunteer individuals of similar age and sex to patients
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
2 Minutes Walking Test | baseline
  Two Minute Walk Test (2MWT) will be performed to evaluate functional mobility.
Timed Up and Go Test | baseline
  Timed Up and Go Test will be performed to evaluate functional mobility.

SECONDARY OUTCOMES:
Respiratory Functions Test | baseline
  Challenging vital capacity (FVC), forced expiratory volume in one second (FEV₁), forced expiratory volume in one second to forced vital capacity (FEV₁/FVC), peak flow rate (PEF), forced vital capacity 25-75% speed (FEF25-75%) will be measured by portable spirometry (Spirolab, Medical International Research, Rome, Italy).
Respiratory Muscle Strength | baseline
  Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) will be measured using portable, electronic, oral pressure measuring device (Micro Medical MicroMPM, UK).
Trunk Impairment Scale | baseline
  Trunk impairment scale assesses static and dynamic sitting balance and trunk coordination. The maximum scores on the static sitting balance, dynamic sitting balance, and coordination subscales are 7, 10, and 6 points, respectively. The total score of Trunk impairment scale ranges between 0 and 23 points, with a higher score representing better trunk control.
Side Bridge Test (core muscles endurance) | baseline
  Subjects were asked to lie on their left or right sides and extend their legs straight. Then the subjects lift their hips off the ground and form a straight line with their bodies. The measurements are recorded with a chronometer as seconds. The tests end when the subjects break the test positions.
Modified Biering-Sorensen test (core muscles endurance) | baseline
  During the test, the subjects are placed in an exercise bed that extends outwardly from the leading edge of the upper body and ensures that the upper iliac spine is flush with the bench edge. Subjects are asked to raise their arms while maintaining body positions.Measurements are recorded in seconds with a stopwatch. The tests will end when the subjects break the test positions.
Trunk Flexion Test (core muscles endurance) | baseline
  Individuals are positioned in such a way that the body is at 60º, knees and hip at a flexion position of 90º. The evaluating physiotherapist supports the feet and fixes the feet on the floor. The measurements are recorded with a chronometer as seconds. The test is terminated when the 60 ° trunk flexion is impaired.
Prone bridge test (core muscles endurance) | baseline
  During the test, the subjects place their elbows on the floor as their starting position and open their feet around the width of their thighs. They keep their body straight without bending over their elbows and toes.The measurements are recorded with a chronometer as seconds. The tests end when the subjects break the test positions.
Sit-ups Test (core muscles power) | baseline
  The test is initiated when the subjects are told "start" and they are asked to flex their upper body up from the floor lifting the lower corner of the scapula from the floor.It is recorded how many times the subjects can perform each test for 30 seconds.
Modified Push-ups Test (core muscles power) | baseline
  In the push-ups test, the subjects are required to push their lower body until their elbows reach a 90° angle. They are then asked to extend their arms straight to return to the starting position.It is recorded how many times the subjects can perform each test for 30 seconds.
Lumbopelvic Stability Test | baseline
  Lumbopelvic stability is assessed using a stabilizer Pressure Biofeedback UnitTM (Chattanooga, Australia). With the participant lying supine on a plinth, the cushion is inflated underneath the participant's lumbar spine to 40 mmHg. Prior to testing, all participants are instructed in the "abdominal hollowing" manoeuvre that activates Transversus Abdominis muscle, and told to perform and continue the contraction this during subsequent lumbopelvic stability testing while attempting to minimize contraction of rectus abdominis. Scores are recorded as the highest level completed (0-5) with a pressure change no greater than 10 mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: MELIKE S CENGİZ, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tzelepis GE, McCool FD. Respiratory dysfunction in multiple sclerosis. Respir Med. 2015 Jun;109(6):671-9. doi: 10.1016/j.rmed.2015.01.018. Epub 2015 Feb 12. PMID 25724874
- [Background] Smeltzer SC, Skurnick JH, Troiano R, Cook SD, Duran W, Lavietes MH. Respiratory function in multiple sclerosis. Utility of clinical assessment of respiratory muscle function. Chest. 1992 Feb;101(2):479-84. doi: 10.1378/chest.101.2.479. PMID 1735276
- [Background] Smeltzer SC, Utell MJ, Rudick RA, Herndon RM. Pulmonary function and dysfunction in multiple sclerosis. Arch Neurol. 1988 Nov;45(11):1245-9. doi: 10.1001/archneur.1988.00520350083020. PMID 3190505
- [Background] Mutluay FK, Gurses HN, Saip S. Effects of multiple sclerosis on respiratory functions. Clin Rehabil. 2005 Jun;19(4):426-32. doi: 10.1191/0269215505cr782oa. PMID 15929512
- [Background] Smeltzer SC, Lavietes MH. Reliability of maximal respiratory pressures in multiple sclerosis. Chest. 1999 Jun;115(6):1546-52. doi: 10.1378/chest.115.6.1546. PMID 10378547
- [Background] Sadovnick AD, Eisen K, Ebers GC, Paty DW. Cause of death in patients attending multiple sclerosis clinics. Neurology. 1991 Aug;41(8):1193-6. doi: 10.1212/wnl.41.8.1193. PMID 1866003
- [Background] Mutluay FK, Demir R, Ozyilmaz S, Caglar AT, Altintas A, Gurses HN. Breathing-enhanced upper extremity exercises for patients with multiple sclerosis. Clin Rehabil. 2007 Jul;21(7):595-602. doi: 10.1177/0269215507075492. PMID 17702701
- [Background] Lanzetta D, Cattaneo D, Pellegatta D, Cardini R. Trunk control in unstable sitting posture during functional activities in healthy subjects and patients with multiple sclerosis. Arch Phys Med Rehabil. 2004 Feb;85(2):279-83. doi: 10.1016/j.apmr.2003.05.004. PMID 14966714
- [Background] Fry DK, Huang M, Rodda BJ. Core muscle strength and endurance measures in ambulatory persons with multiple sclerosis: validity and reliability. Int J Rehabil Res. 2015 Sep;38(3):206-12. doi: 10.1097/MRR.0000000000000109. PMID 25647356
- [Background] Sebastiao E, Sandroff BM, Learmonth YC, Motl RW. Validity of the Timed Up and Go Test as a Measure of Functional Mobility in Persons With Multiple Sclerosis. Arch Phys Med Rehabil. 2016 Jul;97(7):1072-7. doi: 10.1016/j.apmr.2015.12.031. Epub 2016 Mar 2. PMID 26944709
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Black LF, Hyatt RE. Maximal respiratory pressures: normal values and relationship to age and sex. Am Rev Respir Dis. 1969 May;99(5):696-702. doi: 10.1164/arrd.1969.99.5.696. No abstract available. PMID 5772056
- [Background] Standardization of Spirometry, 1994 Update. American Thoracic Society. Am J Respir Crit Care Med. 1995 Sep;152(3):1107-36. doi: 10.1164/ajrccm.152.3.7663792. No abstract available.
- [Background] Verheyden G, Nuyens G, Nieuwboer A, Van Asch P, Ketelaer P, De Weerdt W. Reliability and validity of trunk assessment for people with multiple sclerosis. Phys Ther. 2006 Jan;86(1):66-76. doi: 10.1093/ptj/86.1.66. PMID 16386063
- [Background] Gijbels D, Eijnde BO, Feys P. Comparison of the 2- and 6-minute walk test in multiple sclerosis. Mult Scler. 2011 Oct;17(10):1269-72. doi: 10.1177/1352458511408475. Epub 2011 Jun 3. PMID 21642370
- [Background] Bliss LS, Teeple P. Core stability: the centerpiece of any training program. Curr Sports Med Rep. 2005 Jun;4(3):179-83. doi: 10.1007/s11932-005-0064-y. PMID 15907272
- [Background] Moreau CE, Green BN, Johnson CD, Moreau SR. Isometric back extension endurance tests: a review of the literature. J Manipulative Physiol Ther. 2001 Feb;24(2):110-22. doi: 10.1067/mmt.2001.112563. PMID 11208223
- [Derived] Ozen MS, Calik-Kutukcu E, Salci Y, Karanfil E, Tuncer A, Armutlu K. Is there a relationship between respiratory function and trunk control and functional mobility in patients with relapsing-remitting multiple sclerosis? Neurol Res. 2023 Jul;45(7):619-626. doi: 10.1080/01616412.2023.2176628. Epub 2023 Feb 13. PMID 36780377
- See also: Mills JD, Taunton JE, Mills WA. The effect of a 10-week training regimen on lumbo-pelvic stability and athletic performance in female athletes: a randomized-controlled trial. Physical Therapy in Sport. 2005;6(2):60-6. — https://doi.org/10.1016/j.ptsp.2005.02.006